CLINICAL TRIAL: NCT04698031
Title: Stroke and Coated-Platelets - A Translational Research Initiative
Brief Title: Efficacy of Clopidogrel on Incidence of Silent Brain Infarction
Acronym: ECISBI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NURC-021-20S
Record Dates: First submitted 2020-12-28; First posted 2021-01-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Silent Brain Infarction

STUDY DESIGN:
Intervention Model Description: Patients admitted for stroke/TIA, with indication for antiplatelet therapy as secondary prevention (decision independent of the study and based on individual clinical decision for each patient by the treating physician), will be assigned to therapy with either clopidogrel or aspirin. Both medications are FDA approved for secondary prevention. Patients will be followed for 24 months and repeat brain MRI will be obtained at 24 months. These doses are part of the recommended guidelines for secondary stroke prevention. After randomization, an electronic prescription will be signed by the PI (flagged as part of the research protocol) for a 90-day supply with multiple refills. The medication will be delivered prior to discharge.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The two stroke neurologists reviewing the brain MRI scans will independently adjudicate the presence and number of SBIs for each patient by reviewing the initial and repeat scans, along with the medical history. Each adjudicator will maintain a log with the results and a study identification number while blinded to the platelet procoagulant levels and intervention arm distribution. The laboratory staff will be blinded to clinical, imaging and intervention data. The VA Research Pharmacy will dispense similar looking pills to ensure the double-blind nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clopidogrel (Experimental): After randomization, patients will receive clopidogrel mg daily for the duration of the study. The VA Research Pharmacy will dispense similar looking pills (using a "dummy pill") with Arm 2 to ensure the double-blind nature of the intervention. Clopidogrel is FDA approved for secondary prevention of stroke. Patients will be followed for 24 months with repeat brain MRI scans obtained at 24 months.
  Interventions: Drug: Clopidogrel treatment
- Aspirin (Experimental): After randomization, patients will receive aspirin daily for the duration of the study. The VA Research Pharmacy will dispense similar looking pills (using a "dummy pill") with Arm 1 to ensure the double-blind nature of the intervention. Aspirin is FDA approved for secondary prevention of stroke. Patients will be followed for 24 months with repeat brain MRI scans obtained at 24 months.
  Interventions: Drug: Aspirin treatment

INTERVENTIONS:
Drug: Clopidogrel treatment — After randomization, patients will receive clopidogrel 75 mg daily for the duration of the study. The VA Research Pharmacy will dispense similar looking medication with Arm 2 to ensure the double-blind nature of the intervention. Clopidogrel is FDA approved for secondary prevention of stroke. Follow-up will be for 24 months with repeat brain MRI obtained at 24 months to assess for interval presence of silent brain infarctions.
  Arms: Clopidogrel
Drug: Aspirin treatment — After randomization, patients will receive Aspirin 325 mg daily for the duration of the study. The VA Research Pharmacy will dispense similar looking medication with Arm 2 to ensure the double-blind nature of the intervention. Aspirin is FDA approved for secondary prevention of stroke. Follow-up will be for 24 months with repeat brain MRI obtained at 24 months to assess for interval presence of silent brain infarctions.
  Arms: Aspirin

SUMMARY:
Silent brain infarctions (SBIs) are a manifestation of covert cerebrovascular disease, without obvious clinical deficit, noted very often in patients presenting with a new stroke or new transient ischemic attack. SBIs are linked to a significant increase in risk for subsequent stroke and cognitive decline. However, no biomarker is currently available that can predict the recurrence of these subclinical lesions. Coated-platelets are a measure of platelet procoagulant potential significantly increased in patients with ischemic stroke or transient ischemic attack compared to unaffected controls. Higher coated-platelet levels are strongly associated with both the presence and number of SBIs. Among medications approved for preventing stroke recurrence, we identified clopidogrel as a pharmacological agent leading to a decrease in coated-platelet levels. In this project, we plan to evaluate if clopidogrel can decrease the rate of occurrence of new silent brain infarctions. The result will enhance the investigators understanding of the relationship between platelets and silent brain infarcts, leading to improved health care delivery and also potential targets for novel preventive pharmacological interventions.

DETAILED DESCRIPTION:
Introduction:

Silent brain infarcts (SBIs) are a recently recognized, commonly noted and yet poorly understood finding of cerebral infarction on imaging studies without a clinically apparent neurological deficit. The availability of high resolution brain imaging such as MRI has made the recognition and characterization of these covert markers of cerebrovascular disease possible. SBIs, also referred to as silent strokes, are subcortical cavities or cortical areas of gliosis presumed to be caused by previous infarction.

The prevalence of SBIs in the general population ranges between 8 and 28% in large cardiovascular and aging studies performed in Europe and North America. A key finding has been that prevalence rates are relatively low before age 65 with a gradual increase seen with aging. Among vascular risk factors, hypertension has the strongest association with SBIs, however other vascular risk factors, such as stroke, have been associated with increased prevalence of these lesions. The overall prevalence of SBI far exceeds that of symptomatic stroke and is estimated that for every symptomatic stroke there are approximately 10 SBIs.

Incidence data for SBIs are sparse, likely a reflection of the need for repeat imaging studies. Incidence in the general population is estimated at 3% and 6.5% per year from large population studies. A high incidence of SBIs has been reported following procedures such as aortic valve replacement or carotid endarterectomy, likely directly related to these procedures. Research data in a cohort of TIA patients who underwent initial MRI at the time of the diagnosis and then repeat brain MRI one year after the index event showed a 37% incidence of new SBIs.

There has been considerable evidence linking SBIs with an increased risk for subsequent occurrence of stroke, development of cognitive decline and mortality, suggesting that SBIs are precursors of more severe ischemic brain disease.

Coated-platelets are a class of activated platelets, detected only after simultaneous stimulation with two agonists, thrombin and collagen, or thrombin and convulxin, a collagen receptor agonist from tropical rattlesnake venom. In stroke-free controls, coated-platelets represent approx. 30% of all platelets. Coated-platelet levels are increased in stroke patients as compared to those with lacunar stroke or controls; higher coated-platelet levels measured at the time of the clinical infarct correlate with an increased risk for recurrence at 12 months while lower coated-platelet levels are related to the occurrence of very early inpatient major hemorrhagic complications. These data support a role for platelet procoagulant potential in the balance between thrombosis and hemorrhage.

Several investigations highlight the possibility that coated-platelets play a role in the events preceding stroke. In asymptomatic carotid stenosis, patients with coated-platelet levels 45.2% are at highest risk for incident stroke as compared to those with levels < 45.2 %. In SAH patients, delayed cerebral ischemia (ischemic strokes occurring days after the initial hemorrhage) was linked to a steep increase in coated-platelet levels immediately predating the infarct. Recent work in stroke patients found higher coated-platelet levels significantly associated with the presence and number of SBIs.

Longitudinal data in stroke patients exploring the impact of medications used for secondary stroke prevention identified clopidogrel as the only pharmacological agent leading to a sustained decrease in coated-platelet levels after initiation of therapy. Aspirin, anticoagulation therapy or statins did not lead to a similar effect.

Methods:

The goal of the investigators study is to evaluate the efficacy of clopidogrel on the incidence of silent brain infarction in patients with stroke/TIA using a randomized, double-blind aspirin-controlled clinical trial. The investigator's hypothesis is that clopidogrel treatment will lead to decreased incidence of SBIs in patients with non-lacunar stroke/TIA treated over a two-year period.

Consecutive eligible patients admitted with ischemic stroke or TIA to the Neurology service qualifying for the study (see inclusion and exclusion criteria separately) will be randomized to either clopidogrel or aspirin, stratified by sex. The study statisticians will create the randomization sequence using randomly chosen block sizes of four or six and will implement the sequence concealment. These doses are part of the recommended guidelines for secondary stroke prevention and both medications are FDA approved for secondary stroke prevention.

All patients will be followed by the research team in conjunction with regularly scheduled outpatient visits for up to one year independent of the current study. After the 12-month time point, the investigators will maintain phone contact with each patient for an additional 12 months to decrease loss to follow-up. Prior to the 24-month time point, the PI/Research Assistant will order a repeat non-contrast MRI for each patient.

Initial and repeat MRI images will be independently reviewed after the repeat scan is completed at 24 months by two experienced stroke specialists while blinded to the coated-platelet levels and treatment arm. The initial and repeat MRI will be compared for the presence of new (interval) SBIs in order to determine SBI incidence.

SBIs will be identified on MRI studies, using a 1.5 Tesla magnet, based on published guidelines as focal (ovoid or irregularly shaped), 3mm, cavitary lesions, displaying T1 hypointensity and T2 hyperintensity features, and hypointense on FLAIR sequences. In addition, the cortical SBIs (10% of lesions) may also display some focal atrophic changes of the cerebral cortex in the area surrounding the infarct. These lesions have a chronic appearance, can be easily distinguished from acute ischemic changes through the use of DWI and ADC images and have no corresponding, clinically apparent, cerebrovascular ischemic event noted in the patient's history.

Using electronic medical records, the investigators will collect the following data: prescription medicines, age, sex, race, ethnicity, past medical history, type of stroke, National Institutes of Health Stroke Scale (NIHSS) score upon admission, results of diagnostic studies performed for stroke, vascular risk factors (diabetes, hypertension, large-artery artery disease, atrial fibrillation, prior stroke/TIA, hypercholesterolemia, obesity, cardiac disease, aortic arch plaque, smoking, alcohol consumption), hematological parameters (total platelet count, mean platelet volume, white blood cell count and hemoglobin), and coagulation studies (PT, PTT and INR).

Because prior research linked interval development of SBIs with decline in cognitive function, patients will be screened for cognitive impairment at discharge using the MoCA test. Those with abnormal MoCA results (<26/30 points) will be referred to the Memory Loss clinic for memory loss assessment, including neuropsychological testing. At the end to the follow-up period repeat neuropsychological testing will be performed in individuals who were evaluated initially and compared to the initial results. The investigators will also repeat cognitive screening with MOCA in patients who scored within normal range initially, and those with abnormal results at 24 months will undergo memory loss assessment.

Statistical analysis:

A target sample size of 152 participants (76 clopidogrel and 76 aspirin) over 1.5 years (8.4 patients/month) is sufficient to provide preliminary estimates of the effect size and variation in efficacy, as well as feasibility information regarding the conduct of the clinical trial. This calculation provides 80% power to detect a 65% reduction in the hazard of SBI for those receiving clopidogrel versus aspirin, assuming a 2-sided 0.05 alpha level, loss-to-follow-up and death rates of 10%, and follow-up for 24 months. Even if the effect size observed in the clinical trial is not as large, the trial will still generate valuable estimates of effect size and variation for efficacy, as well as feasibility information. These estimates can be used to design a larger, more definitive clinical trial.

The time to incident SBI distribution will be compared between the clopidogrel and aspirin arms using a log-rank test. Adverse event will be compared between the treatment groups using a Chi-square test, or Fisher's exact test for rare events. Analyses will be based on the intention-to-treat principle. A separate per-protocol analysis, analyzing data from all patients who adhered to the study medication will be performed. No formal interim efficacy analyses will be performed. Data quality, protocol implementation, retention and patient adherence and adverse events will be summarized every six months. Statistical significance will be set at p<0.05. A multiple imputation method will be used to impute missing data.

Anticipated findings:

The investigators anticipate that treatment with clopidogrel at standard dose for secondary stroke prevention will lead to a significant decrease in the incidence of SBIs as compared to treatment with aspirin. The current data will provide proof of concept for future larger trials with more extended follow-up time that are able to also evaluate reduction on key cardiovascular outcomes, such as stroke, myocardial infarction and sudden death. In addition, key data regarding clinical and imaging features of patients with SBI and progression of cognitive impairment will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ischemic stroke/TIA
* < 90 days from onset of symptoms
* initial MRI available,
* not receiving antiplatelet therapy at the time of admission
* medical decision by the treating physician that antiplatelet therapy is indicated for secondary prevention (decision independent of the study and based on individual clinical decision for each patient).
* baseline coated-platelet levels at 40%,
* willingness to participate in the study for 24 months

Exclusion Criteria:

* dementia (based on chart review or self/proxy report)
* > 90 days from onset of symptoms
* initiation of anticoagulation or thrombolytics prior to phlebotomy
* intracranial hemorrhage or bleeding diatheses
* end-stage renal disease (ESRD)
* inability to tolerate consenting or phlebotomy
* prior adverse/allergic reactions to clopidogrel
* treating physician deemed a different antiplatelet dose or dual antiplatelet therapy as the only treatment choice

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
new silent brain infarctions | 24 months
  Each of the two reviewers will independently adjudicate the presence, location and number of SBIs for each patient by reviewing both the initial and repeat scans at 24 months.

SECONDARY OUTCOMES:
cognitive impairment | 24 months
  The presence and severity of cognitive impairment will be assessed at the end of the follow-up period (24 months) using the Montreal Cognitive Assessment (MoCA) test. Patients with abnormal results (MoCA test score < 26/30) will undergo memory loss assessment in the VA Memory Loss clinic . The assessment will include neuropsychological testing, serology studies, and additional neuroimaging, if indicated, in accordance with published guidelines. All patients will be classified initially into one of two categories: 1) presence of cognitive impairment or 2) no cognitive impairment. Patients with cognitive impairment will be subsequently subcategorized after their clinic evaluation into 1) MCI [Clinical Dementia Rating (CDR) = 0.5] or 2) dementia (CDR > 0.5).

CONTACTS AND LOCATIONS:
Overall Officials: Calin Ioan Prodan, MD, Principal Investigator — Oklahoma City VA Medical Center, Oklahoma City, OK
Locations (1):
- Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwan J, Hafdi M, Chiang LLW, Myint PK, Wong LS, Quinn TJ. Antithrombotic therapy to prevent cognitive decline in people with small vessel disease on neuroimaging but without dementia. Cochrane Database Syst Rev. 2022 Jul 14;7(7):CD012269. doi: 10.1002/14651858.CD012269.pub2. PMID 35833913